CLINICAL TRIAL: NCT04643067
Title: A Phase 1b/2a Multicenter Study to Assess the Safety and Tolerability, Pharmacokinetics, and Preliminary Efficacy of KPG-818 in Patients With Systemic Lupus Erythematosus
Brief Title: Phase 1b/2a Study to Evaluate Safety and Efficacy of KPG-818 in SLE
Acronym: Lupus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kangpu Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPG-818-SLE
Record Dates: First submitted 2020-11-12; First posted 2020-11-24 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: SLE; Drug
MeSH Terms: conditions — drug-induced lupus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KPG-818 low dose (Active Comparator): After providing informed consent, patients will be assessed for study eligibility at the Screening visit. A total of 8 to 12 patients will be randomized to receive this dose level of KPG-818 in a double-blind fashion. Patients will receive treatment for 12 weeks with a 4-week safety follow-up. Capsules of this level of dosage will be taken orally in the morning once a day. All patients will return for follow-up visits after their final dose. The total duration of study participation for each patient (from Screening through Follow-up visit) is anticipated to be approximately 20 weeks.
  Interventions: Drug: KPG-818 low dose
- KPG-818 mid dose (Active Comparator): After providing informed consent, patients will be assessed for study eligibility at the Screening visit. A total of 8 to 12 patients will be randomized to receive this dose level of KPG-818 in a double-blind fashion. Patients will receive treatment for 12 weeks with a 4-week safety follow-up. Capsules of this level of dosage will be taken orally in the morning once a day. All patients will return for follow-up visits after their final dose. The total duration of study participation for each patient (from Screening through Follow-up visit) is anticipated to be approximately 20 weeks.
  Interventions: Drug: KPG-818 mid dose
- KPG-818 high dose (Active Comparator): After providing informed consent, patients will be assessed for study eligibility at the Screening visit. A total of 8 to 12 patients will be randomized to receive this dose level of KPG-818 in a double-blind fashion. Patients will receive treatment for 12 weeks with a 4-week safety follow-up. Capsules of this level of dosage will be taken orally in the morning once a day. All patients will return for follow-up visits after their final dose. The total duration of study participation for each patient (from Screening through Follow-up visit) is anticipated to be approximately 20 weeks.
  Interventions: Drug: KPG-818 high dose
- Placebo arm (Placebo Comparator): After providing informed consent, patients will be assessed for study eligibility at the Screening visit. A total of 8 to 12 patients will be randomized to receive this dose level of KPG-818 in a double-blind fashion. Patients will receive treatment for 12 weeks with a 4-week safety follow-up. Capsules of this level of dosage will be taken orally in the morning once a day. All patients will return for follow-up visits after their final dose. The total duration of study participation for each patient (from Screening through Follow-up visit) is anticipated to be approximately 20 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KPG-818 low dose — The dose levels may be modified according to the results from phase 1b of the study. Dose adjustment is allowed during the study.
  Arms: KPG-818 low dose
Drug: KPG-818 mid dose — The dose levels may be modified according to the results from phase 1b of the study. Dose adjustment is allowed during the study.
  Arms: KPG-818 mid dose
Drug: KPG-818 high dose — The dose levels may be modified according to the results from phase 1b of the study. Dose adjustment is allowed during the study.
  Arms: KPG-818 high dose
Drug: Placebo — This is the comparative arm.
  Arms: Placebo arm

SUMMARY:
Study Title

A phase 1b/2a multicenter, randomized, double-blind, placebo-controlled study to assess the safety and tolerability, pharmacokinetics and preliminary efficacy of KPG-818 in patients with mild to moderate systemic lupus erythematosus

DETAILED DESCRIPTION:
This is a Phase 1b/2a multicenter study to evaluate the safety, PK, PD, and clinical efficacy of KPG-818 in patients with SLE. The trial will consist of 2 parts: Phase 1b, a multiple-ascending dose (MAD) study; and Phase 2a, a proof of concept (POC) study.

ELIGIBILITY:
Inclusion criteria are listed as follows:

1. Age≥18
2. BMI between 18-40kg/m²
3. Diagnosed with SLE according to the 2019 EULAR/ACR criteria for SLE
4. Meeting SLE activity requirements
5. Males and females childbearing potential must agree to use contraception methods
6. All patients must:

   1. Understand that KPG-818 could have potential teratogenic risk.
   2. Agree not to share KPG-818 with another person.
   3. Be counseled about pregnancy precautions and risks of fetal exposure as described in the Pregnancy Prevention Plan.
7. Patients must agree not to donate blood (or any component of blood) from 3 months before Screening until 3 months after the last dose of KPG-818.
8. Patients must be willing to comply with precautions to reduce the risk of COVID-19 infection and to undergo COVID-19 PCR test.

Exclusion criteria are listed as follows:

1. Use of any prohibited medications within the pre-specified time
2. Patients must meet exclusionary lab criteria
3. Active and/or unstable neuropsychiatric SLE
4. Active or history of severe systemic bacterial, viral, fungal, mycobacterial, or parasitic infections within 6 months prior to Screening
5. Current or recent sign or symptoms of infections, or severe viral infections
6. Conditions predisposes patient to infection
7. Active TB or positive QuantiFERON®-TB Gold test
8. Patients with malignancy and antiphospholipid syndrome history
9. Inflammatory joint or skin disease, mixed connective tissue disease, scleroderma, and/or overlap syndromes, or acute or chronic disease
10. Concomitant condition that required systemic corticosteroid use within 1 year before Screening
11. Alcohol or drug abuse history
12. Positive urine drug test at screening
13. History or planned major surgery
14. Pregnant or breastfeeding female
15. Signs or symptoms of COVID-19 infection
16. Known allergic reaction to any of the ingredients for study drug or placebo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Safety assessment by the occurrence of adverse events (AEs) | 4 weeks for phase Ib and 16 weeks for phase IIa
  To calculate the occurrence rate of adverse events (AEs)
Safety assessment by the changes from baseline in laboratory parameters | 4 weeks for phase Ib and 16 weeks for phase IIa
  To calculate the occurrence rate of out of normal ranges of laboratory parameter changes from baseline.
Safety assessment by out of normal range of vital signs | 4 weeks for phase Ib and 16 weeks for phase IIa
  To calculate the occurrence rate of out of normal range of vital signs from baseline.
Safety assessment by out of normal range of ECG results | 4 weeks for phase Ib and 16 weeks for phase IIa
  To calculate the occurrence rate of out of normal range of ECG results.
PK profile of time to peak (Tmax) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured on Day 1 after dose administration and after the plasma concentration reaches a steady state.
PK profile of peak plasma concentration (Cmax) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured on Day 1 after dose administration.
PK profile of elimination half-life (t1/2) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured on Day 1 after dose administration and after the plasma concentration reaches a steady state.
PK profile of the area under the concentration-time curve (AUC0-24h) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured on Day 1 after dose administration.
PK profile of the mean retention time (MRT) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured after the plasma concentration reaches a steady state.
PK profile of trough concentrations at steady state (Css_min) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured after the plasma concentration reaches a steady state.
PK profile of peak concentrations at steady state (Css_max) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured after the plasma concentration reaches a steady state.
PK profile of the area under the concentration-time curve at steady state (AUCτ, AUC0-∞) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured after the plasma concentration reaches a steady state.
PK profile of the clearance (CL/F) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured after the plasma concentration reaches a steady state.
PK profile of the apparent volume of distribution ((Vz/F) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured after the plasma concentration reaches a steady state.
PK profile of the cumulative coefficient (R) for KPG-818 and KPG-818H (if applicable). | 4 weeks for phase Ib and 16 weeks for phase IIa
  This will be measured after the plasma concentration reaches a steady state.
Assess the proportion of patients with improvement of clinical scores of SELENA-SLEDAI (safety of estrogens in lupus national assessment-systemic lupus erythematosus disease activity index) improvement ≥ 4 points from baseline at Week 12. | 16 weeks for phase IIa
  To calculate the proportion of patients with SELENA-SLEDAI (safety of estrogens in lupus national assessment-systemic lupus erythematosus disease activity index) improvement ≥ 4 points from baseline at Week 12. Note: the SELENA-SLEDAI scale ranges from 0~105, with 105 as the highest disease activity.

SECONDARY OUTCOMES:
Mean change from baseline in PGA (Physician Global Assessment) score at Week 12. | 16 weeks for phase IIa
  Mean change from baseline in PGA (Physician Global Assessment) score at Week 12. Note: the PGA is a visual scale for the physician to mark, from 0mm to 100mm, with 0mm being no disease activity and 100mm being the extreme disease activity.
The proportion of patients with a ≥ 50% reduction from baseline in CLASI (Cutaneous Lupus erythematosus disease Area and Severity Index) activity score at Week 12, in patients with baseline CLASI activity score ≥ 10. | 16 weeks for phase IIa
  The proportion of patients with a ≥ 50% reduction from baseline in CLASI (Cutaneous Lupus erythematosus disease Area and Severity Index) activity score at Week 12, in patients with baseline CLASI activity score ≥ 10. Note: the total CLASI score ranges from 0 to 114, with 0 being the least disease activity and 114 being the most.
Number of patients with adverse event at Week 12 | 12 weeks for phase IIa
  Number of patients with adverse event at Week 12
Number of patients with adverse event at Week 16. | 16 weeks for phase IIa
  Number of patients with adverse event at Week 16.
The PK endpoint of the measurement of area under the curve (AUC) at Week 12 (AUC0-last) for assessment of KPG-818 and KPG-818H (if applicable). | 12 weeks for phase IIa
  The PK endpoint of the measurement of area under the curve (AUC) at Week 12 (AUC0-last) for assessment of KPG-818 and KPG-818H (if applicable).
The PK endpoint of the maximum observed concentration (Cmax) at Week 12 for assessment of KPG-818 and KPG-818H (if applicable) | 12 weeks for phase IIa
  The PK endpoint of the maximum observed concentration (Cmax) at Week 12 for assessment of KPG-818 and KPG-818H (if applicable)
The PK endpoint of time to Cmax (tmax) at Week 12 for assessment of KPG-818 and KPG-818H (if applicable) | 12 weeks for phase IIa
  The PK endpoint of time to Cmax (tmax) at Week 12 for assessment of KPG-818 and KPG-818H (if applicable).
The PK endpoint of Ctrough throughout the dosing period for assessment of KPG-818 and KPG-818H (if applicable) | 12 weeks for phase IIa
  The PK endpoint of Ctrough throughout the dosing period for assessment of KPG-818 and KPG-818H (if applicable)
The PK endpoint of serum concentrations by scheduled timepoints for assessment of KPG-818 and KPG-818H (if applicable) | 12 weeks for phase IIa
  The PK endpoint of serum concentrations by scheduled timepoints for assessment of KPG-818 and KPG-818H (if applicable)

OTHER OUTCOMES:
Explore the mean change from baseline in potential biomarker, i.e. Aiolos, of KPG-818 in PBMCs and CD19+ B Cells at Week 2. | 2 weeks for phase Ib
  Explore the mean change from baseline in potential biomarker of Aiolos of KPG-818 in PBMCs and CD19+ B Cells at Week 2.
Explore the mean change from baseline in potential biomarker, i.e. Ikaros, of KPG-818 in PBMCs and CD19+ B Cells at Week 2. | 2 weeks for phase Ib
  Explore the mean change from baseline in potential biomarker, i.e. Ikaros, of KPG-818 in PBMCs and CD19+ B Cells at Week 2.
Explore the mean change from baseline in potential biomarker, i.e. CRBN proteins, of KPG-818 in PBMCs and CD19+ B Cells at Week 2. | 2 weeks for phase Ib
  Explore the mean change from baseline in potential biomarker, i.e. CRBN proteins, of KPG-818 in PBMCs and CD19+ B Cells at Week 2.
Mean change from baseline in potential biomarker, i.e. CRBN proteins, of KPG-818 in PBMCs and CD19+ B cells at week 12 | 12 weeks for phase IIa
  Mean change from baseline in potential biomarker, i.e. CRBN proteins, of KPG-818 in PBMCs and CD19+ B cells at week 12
Mean change from baseline in potential biomarker, i.e. Aiolos, of KPG-818 in PBMCs and CD19+ B cells at week 12 | 12 weeks for phase IIa
  Mean change from baseline in potential biomarker, i.e. Aiolos, of KPG-818 in PBMCs and CD19+ B cells at week 12
Mean change from baseline in potential biomarker, i.e. Ikaros, of KPG-818 in PBMCs and CD19+ B cells at week 12 | 12 weeks for phase IIa
  Mean change from baseline in potential biomarker, i.e. Ikaros, of KPG-818 in PBMCs and CD19+ B cells at week 12
Mean change from baseline in absolute counts of CD 19+ B cell and CD3+ T cell at week 12 | 12 weeks for phase IIa
  Mean change from baseline in absolute counts of CD 19+ B cell and CD3+ T cell at week 12
Mean change from baseline in IgA, IgG and IgM in serum at week 12 | 12 weeks for phase IIa
  Mean change from baseline in IgA, IgG and IgM in serum at week 12
Dose regimens for a Phase 2b/phase 3 study | 4 weeks for phase Ib and 16 weeks for phase IIa
  Dose regimens for a Phase 2b/phase 3 study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Kangpu Biopharmaceuticals, Ltd.
Locations (18):
- United States (18):
  - Anniston Medical Clinic, Anniston, Alabama
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Hope Clinical Trials, Inc., Coral Gables, Florida
  - JY Research Institute Inc, Cutler Bay, Florida
  - OSIS Clinical Research, Hollywood, Florida
  - SouthCoast Research Center Inc, Miami, Florida
  - D & H National Research Centers, Miami, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Omega Research MetroWest LLC, Orlando, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Oracle Clinical Research, College Park, Georgia
  - STAT Research, Vandalia, Ohio
  - Shelby Research LLC, Memphis, Tennessee
  - Accurate Clinical Management, Houston, Texas
  - Accurate Clinical Research LLC, Houston, Texas
  - Sun Research Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No